CLINICAL TRIAL: NCT02654444
Title: Concordance Study of Her2 Expression Level in Breast Cancer Tissues
Brief Title: Semi-Quantification of Her2/Neu Protein Expression in Formalin Fixed, Paraffin-Embedded Normal and Neoplastic Tissue
Status: Completed | Type: Observational
Sponsor: Applied Spectral Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASI-HER2-IHC
Record Dates: First submitted 2015-02-05; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Immunohistochemical (IHC); Her2/Neu; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- GenASIs HiPath IHC #1: Expression of HER2 antibody. Semi-Quantitative value
- GenASIs HiPath IHC #2: Expression of HER2 antibody. Semi-Quantitative value
- GenASIs HiPath IHC #3: Expression of HER2 antibody. Semi-Quantitative value

SUMMARY:
The purpose of the study is the identification and quantification of protein expression level in breast cancer tissues.

The imaging system is intended for diagnostic use as an aid to the pathologist in the detection, counting and classifying her2 immunohistochemical (IHC) stained samples.

DETAILED DESCRIPTION:
The anti Her2/neu Kit is a semi-quantitative immunohistochemical (IHC) assay to identify the Human Epithelial growth factor receptor (Her2/neu) expression in formalin-fixed, paraffin-embedded human breast cancer tissue specimens. Results from the Her-2 test is indicated as an aid in the assessment of patients for whom HERCEPTIN® (Trastuzumab) treatment is being considered. While the Her-2 kit provides the antibodies that offer direct visualization and semi-quantification of the HER2 protein expression through a brightfield microscope, the GenASIs GoPath system is designed to complement the routine workflow of the pathologist in the review of immunohistochemically stained histologic slides.

ELIGIBILITY:
Inclusion Criteria:

* Women having breast cancer aged 21 and up
* Borders of tumor nuclei are distinguishable
* Nuclei should have good integrity
* Background should not contain particles that interfere with the analysis

Exclusion Criteria:

* Slides that cannot be analyzed manually by Pathologist

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women having breast cancer
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
IVD study of HER2 IHC samples: Accuracy of analysis | 1 Day
  Comparison tests (accuracy) between manual and automatic analysis of antibody expressions. The results from the automatic counting from the clinical studies will be compared to the manual counting analysis.
  The study is declared Success if the lower limit of two-sided 95% exact Binomial confidence interval for I. Positive, Negative and Overall agreement with manual count will be at least 85% II. Equivocal agreement with manual count will be at least 80%
IVD study of HER2 IHC samples: Repeatability & Reproducibility of analysis | 1 Day
  Repeatability & Reproducibility tests of system analysis of antibody expressions. R&R acceptance criteria of HER2 are related to the average agreement for between runs, between days and between systems The R&R part of the study will be declared "Success" based on the two-level HER2/neu outcome (negative=0 & 1+, positive=2+ & 3+), if positive and negative average agreements will be at least 85%